CLINICAL TRIAL: NCT06242054
Title: The Development and Clinical Application of a Motor Function Assessment System Based on Video Tracking and Artificial Intelligence Technique
Brief Title: Motor Function Assessment System Based on Video Tracking and Artificial Intelligence Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Zhou Feifei, Deputy Director of Orthopedics Department, Peking University Third Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: M2021454
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Cervical Spine Myelopathy
Keywords: Cervical spine myelopathy; Hand motor funciton; Video tracking technology; Artificial intelligence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with cervical spine myelopathy (Experimental)
  Interventions: Diagnostic Test: Motor Function Assessment System
- Healthy people (Other)
  Interventions: Diagnostic Test: Motor Function Assessment System

INTERVENTIONS:
Diagnostic Test: Motor Function Assessment System — Participants were instructed to extend their fingers and subsequently clench their fists to the maximum possible range of motion, in order to complete the evaluation of Motor Function Assessment System.

SUMMARY:
The goal of this clinical trial is to develop a motion recognition system based on video tracking technology and combine it with artificial intelligence technology to form a motion recognition and function evaluation system in in healthy people and patients with cervical spondylotic myelopathy. The main questions it aims to answer are:

* The development of this motion recognition system,
* In the scenario of hand motor dysfunction, the key parameters of hand movement in healthy people and patients with cervical spondylotic myelopathy were evaluated, and the hand motor function model was established to achieve an objective, highly sensitive, highly specific, repeatable and easy-to-use system in clinical hand motor function evaluation.

Participants will recieved the evaluation of this system and mJOA before the surgery.

If there is a comparison group: Researchers will compare the evaluation results of healthy people to see if this system could recognized the hand motor dysfunction of patients with cervical spondylotic myelopathy.

ELIGIBILITY:
Inclusion Criteria:

* Study Group: 1. Patients with cervical spondylotic myelopathy diagnosed by clinical symptoms and cervical spine imaging examination (including cervical flexion and extension X-ray, cervical spine CT and cervical spine MRI).
* Control Group: 1. Healthy people without clinical and imaging manifestations of cervical spondylotic myelopathy.
* Age 18-80 years old.
* Can complete the informed consent process.

Exclusion Criteria:

* Patients with hand dysfunction caused by other reasons (such as rheumatoid arthritis, history of hand trauma, history of hand surgery, etc.).
* Patients who cannot complete the assessment process due to various reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Motor Function Assessment System | Before the surgery
  Motor Function Assessment System
mJOA | Before the surgery
  mJOA
10-Seconds Grab and Release Test | Before the surgery
  10-Seconds Grab and Release Test

CONTACTS AND LOCATIONS:
Locations (1):
- Feifei Zhou, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No